CLINICAL TRIAL: NCT05903352
Title: Customized Antibiotic Treatment Duration Among Hospitalized Patients With Moderately Severe Community-Acquired Pneumonia
Acronym: CAT-CAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220814; 2023-504208-27-00 (Other: EU CT number)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Community-Acquired Pneumonia
Keywords: Community-Acquired Pneumonia; Antibiotic treatment duration; Antibiotic resistance; Infectious diseases
MeSH Terms: conditions — Community-Acquired Pneumonia; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: All eligible patients with confirmed CAP and willing to participate will be included and randomly assigned (1:1 ratio) by the investigator, to either continue the antimicrobial treatment for a duration predetermined by the investigator (usual practice, at least 3 days of treatment in total), or to stop the antibiotic treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment (Placebo Comparator): Antibiotic treatment duration left to the physician's judgment (usual practice: total treatment duration between 5 to 10 days according to French guidelines; more than 7 days of treatment should be justified).
  Interventions: Drug: Continue the antimicrobial treatment
- Interruption of treatment (Experimental): Interruption of treatment based on the patient reaching all of the following stability criteria (body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure > 90mmHg; oxygen saturation ≥ 92%; respiratory rate < 24/min; normal mental status (27)), with a treatment duration no shorter than 48 h.
  Interventions: Other: Stop antibiotic

INTERVENTIONS:
Other: Stop antibiotic — Stop the antibiotic treatment on day S (stability criteria reached for 24 h or within 48 hours after the start of antibiotic treatment).
  Arms: Interruption of treatment
Drug: Continue the antimicrobial treatment — Continue the antimicrobial treatment for a duration predetermined by the investigator (usual practice, at least 5 days of treatment in total).
  Arms: Antibiotic treatment

SUMMARY:
The primary objective of the study is to evaluate if the efficacy of an experimental strategy on antibiotic treatment duration based on stopping treatment when stability criteria are reached after at least 48 h of treatment, is non-inferior to the efficacy of standard antibiotic duration in CAP patients treated in the hospital setting.

As the secondary objectives, the study aims

* To study if the efficacy of our experimental strategy on antibiotic treatment duration compared to standard of care in CAP patients treated in the hospital setting is non-inferior in terms of:

  * Persistence of cure at Day 30 of antibiotic treatment
  * All-cause mortality rate on Day 30 of antibiotic treatment
  * Patients evolution of pneumonia symptoms and quality of life via 2 scores (CAP score, CAP Sym) at Day 0 of treatment (retrospectively), at stability (Day S), at Day 7 , at Day 15, and at Day 30 of antibiotic treatment.
* To compare between the 2 study arms at Day 30 of antibiotic treatment:

  * The duration of antibiotic treatment;
  * The length of hospital stay;
  * The frequency and severity of adverse events during the 30 days after the start of treatment.
* To explore the impact of reduced antibiotic treatment duration for CAP on the oropharyngeal resistome.

DETAILED DESCRIPTION:
Recent studies have suggested that community-acquired pneumonia (CAP) can be successfully treated with short-course antibiotic regimen when clinical improvement is rapidly obtained. Even if clinical response is obtained in 3 days in the majority of cases, it can vary widely among patients suggesting "one duration does not fit all". An individualised duration of therapy depending on the patient's response could help to ensure bacterial eradication while avoiding unnecessary antibiotic exposure and thus reduce antibiotic resistance. At present, this strategy has never been tested.

This is a phase III, pragmatic, non-inferiority randomised (1:1) national multicentre trial. Population of study participants will be patients admitted to hospital with suspected CAP and in need for antibiotics.

There is no need to establish a DSMB for this trial. The antibiotic treatments prescribed during this study are treatments used in current practice, with well-known adverse drug reactions. Furthermore, a 3-day treatment duration has already been studied in 2 previous randomized clinical trials, showing its safety for hospitalized CAP.

Statistical analysis:

Statistical inference for non-inferiority will be based on the confidence intervals (CI) of the difference in Day 15 cure proportions [proportion in reference arm - proportion in experimental arm] accounting for randomisation stratification factors (centre and delay from Day 0 to Day S (≤ 3 days or > 3 days).

The inferiority hypothesis will be rejected and non-inferiority will be claimed if the upper bound of the 95%CI of the difference is ≤ 10%.

Secondary efficacy endpoints evaluating the evolution of symptoms will be analysed using either a GMM or a GEE for categorical and continuous variables, respectively.

Other quantitative variables will be compared using the Student t-test (or a non-parametric test if the distribution remains skewed following transformation), while categorical variables will be analysed using either the Chi-squared or the Fisher-exact tests.

All statistical tests will be performed with a level of significance of 5%, except the primary endpoint which be analysed with a 2.5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Admitted to hospital for suspected CAP defined by the presence of at least 2 of the following diagnostic clinical criteria:

  * Fever (temperature > 38°C) or hypothermia (< 36°C)
  * Dyspnea
  * Cough
  * Production of purulent sputum
  * Crackles
* Radiological evidence of a new infiltrate (chest X-ray or CT scan)
* Negative viral respiratory testing
* Treated for a minimum of 48 hours with antibiotics (excluding azithromycin due to its prolonged half-life)Presenting with an early clinical response within the last 24 hours (up to 7 days after the start of antibiotic treatment, if planned treatment duration > 7 days), defined by the presence of all the following criteria:apyrexia (T°C ≤ 37.8)heart rate < 100/minrespiratory rate < 24/min, according to the patient's usual mode of oxygenation,arterial oxygen saturation ≥ 92%, according to the patient's usual mode of oxygenation,Patient currently under antibiotic treatment for his suspected CAP (i.e. the last dose of ATB has been administered to the patient less than 24 hours ago)
* Patient presenting a clinical response within the last 24 hours defined by the presence of all the following criteria:

  * apyrexia (T°C ≤ 37.8)
  * heart rate < 100/min
  * respiratory rate < 24/min, according to the patient's usual mode of oxygenation,
  * arterial oxygen saturation ≥ 92%, according to the patient's usual mode of oxygenation,
  * systolic blood pressure ≥ 90mmHg, The last occurring of these criteria must have appeared within the last 24 hours.
* The antibiotic treatment for suspected CAP has started at least 48 hours ago and at most 6 days ago
* No other site of infection besides respiratory
* Affiliated to Health insurance
* Has given informed consent
* Patient understanding oral and written French, or presence of a relative who can explain and help him complete the study documents

Exclusion Criteria:

* Signs of severe CAP (abscess, massive pleural effusion, serious chronic respiratory insufficiency)
* Known immunosuppression (asplenia, neutropenia, agammaglobulinemia, transplant, myeloma, lymphoma, known HIV and CD4<200/mm3)
* Suspected or confirmed legionellosis
* Any other infection necessitating concomitant antibiotic treatment
* Confirmed or suspected aspiration pneumonia or healthcare-associated pneumonia
* Treatment of suspected CAP with azithromycin (due to its prolonged half-life)
* Concomitant steroid treatment (only for patients treated with fluoroquinolones antibiotics)
* Pre-existing aortic aneurysm or dissection, family history of aortic aneurysm or dissection, Marfan syndrome, Ehlers-Danlos syndrome, Takayasu arthritis, uncontrolled arterial hypertension, atherosclerosis (only for patients treated with fluoroquinolones antibiotics)
* Pregnant or breastfeeding woman
* Life expectancy < 1 month
* Patient under legal guardianship (French "tutelle" or "curatelle")
* Patient without fixed address
* Patient enrolled in another interventional clinical trial on CAP treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate of cure at Day 15 after treatment initiation | Day 15
  Cure at Day 15 will be defined by the association of:
  * Persistence of stability criteria (body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure > 90mmHg; oxygen saturation ≥ 92%; respiratory rate < 24/min; normal mental status);
  * No additional antibiotic treatment, targeting CAP, taken after the end of initial antibiotic treatment.
  Patients who died, or are not cured as defined above, will be classified as failure at Day 15.

SECONDARY OUTCOMES:
Rate of cure at Day 30 | Day 30
  Rate of cure at Day 30 after the start of treatment defined by the association of: persistence of stability criteria (body temperature ≤ 37.8°C; heart rate ≤ 100/min; systolic blood pressure > 90mmHg; O2 saturation ≥ 92%; respiratory rate < 24/min; normal mental status); absence of additional antibiotic treatment needed after the end of initial antibiotic treatment.
Mortality on Day 30 | Day 30
  All-cause mortality on Day 30 after the start of antibiotic treatment.
Patients' evolution of pneumonia symptoms | Day-0, Day S, Day 7, at Day 15, and at Day 30
  Patients' evolution of pneumonia symptoms by CAP Score at Day 0 of treatment (retrospectively), at stability (Day S), at Day 7, at Day 15, and at Day 30 of antibiotic treatment.
Patients' evolution of pneumonia symptoms | Day 15 and Day 30
  Patients' evolution of pneumonia symptoms and quality of life by CAP Sym:
  validated self-questionnaires filled at Day 0 of treatment (retrospectively), at stability (Day S), at Day 7, at Day 15, and at Day 30 of antibiotic treatment.
Duration of antibiotic treatment targeting CAP | Day 30
  Duration of antibiotic treatment targeting CAP during the 30 days after the start of treatment.
Duration of antibiotic treatment for all indications | Day 30
  Duration of antibiotic treatment for all indications during the 30 days after the start of treatment.
Length of hospitalization | Day 30
  Length of initial hospital stay
Incidence of adverse event | Day 30
  Frequency and severity of adverse events during the 30 days after the start of treatment
Number of resistance genes | Day S and Day 30
  Calculating for each patient, the number of resistance genes normalised against the quantity of total bacterial DNA, the bacterial richness and diversity, among 300 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Dihn, MD, PhD, Principal Investigator — Infectious diseases department, Raymond-Poincaré Hospital - APHP; Jacques Ropers, PharmD, Study Director — Clinical Research Unit Pitié Salpêtrière - Charles Foix, CHU La Pitié-Salpêtrière - APHP
Locations (1):
- Infectious diseases department, Raymond-Poincaré Hospital - APHP, Garches, France

REFERENCES:
- [Background] Dinh A, Ropers J, Duran C, Davido B, Deconinck L, Matt M, Senard O, Lagrange A, Makhloufi S, Mellon G, de Lastours V, Bouchand F, Mathieu E, Kahn JE, Rouveix E, Grenet J, Dumoulin J, Chinet T, Pepin M, Delcey V, Diamantis S, Benhamou D, Vitrat V, Dombret MC, Renaud B, Perronne C, Claessens YE, Labarere J, Bedos JP, Aegerter P, Cremieux AC; Pneumonia Short Treatment (PTC) Study Group. Discontinuing beta-lactam treatment after 3 days for patients with community-acquired pneumonia in non-critical care wards (PTC): a double-blind, randomised, placebo-controlled, non-inferiority trial. Lancet. 2021 Mar 27;397(10280):1195-1203. doi: 10.1016/S0140-6736(21)00313-5. PMID 33773631